CLINICAL TRIAL: NCT07121764
Title: Comparison of Post-Operative Analgesia With Bupivacaine Alone Versus Bupivacaine and Dexmedetomidine, in Caudal Block for Infra-Umbilical Surgeries in Children
Brief Title: Postoperative Pain Relief in Children: Comparing Caudal Bupivacaine Alone Versus Bupivacaine With Dexmedetomidine for Infra-Umbilical Surgeries Under General Anesthesia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Allama Iqbal Teaching Hospital (Other Government)
Responsible Party: Principal Investigator, Sajid Ullah, Principal Investigator, Allama Iqbal Teaching Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: U1111-1326-5938
Record Dates: First submitted 2025-08-07; First posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Hernia Repair; Orchiopexy; Hypospadias
Keywords: Bupivacaine; Dexmedetomidine; Caudal block; Pediatrics; Postoperative analgesia
MeSH Terms: conditions — Hypospadias | interventions — Dexmedetomidine; Bupivacaine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Monotherapy (Active Comparator): Bupivacaine alone
  Interventions: Drug: Bupivacaine %0.25 (isobaric)
- Combination therapy (Experimental): Bupivacaine with Dexmedetomidine
  Interventions: Drug: Dexmedetomidine & Bupivacaine.

INTERVENTIONS:
Drug: Bupivacaine %0.25 (isobaric) — 1 ml/kg of 0.25% Bupivacaine will be used for caudal block.
  Arms: Monotherapy
Drug: Dexmedetomidine & Bupivacaine. — 1 ml/kg of 0.25% Bupivacaine PLUS 1 μg/kg Dexmedetomidine in 1 ml Normal Saline will be used for caudal block.
  Arms: Combination therapy

SUMMARY:
This study is being done to find out which medicine combination provides better pain relief after surgery in children. Children who are having surgery below the belly button (called infra-umbilical surgery) will receive general anesthesia and a type of pain-blocking injection called a caudal block. This block helps reduce pain after surgery.

The study will compare two types of caudal injections:

One group will receive Bupivacaine alone, a commonly used local anesthetic.

The other group will receive Bupivacaine combined with Dexmedetomidine, a medicine that might help the pain relief last longer.

The main question the researchers want to answer is:

Does adding Dexmedetomidine to Bupivacaine increase the duration of pain relief after surgery in children?

Researchers will also look at:

How long it takes before the child needs the first dose of pain medicine after surgery

How much pain medicine is used in the first 24 hours

How long any movement problems (motor block) last

Whether there are any side effects

Each child will be randomly assigned (like flipping a coin) to one of the two groups. The caudal block will be done after the surgery is completed, while the child is still under anesthesia. The nurse assessing the child's pain will not know which medicine the child received.

Children will be monitored for pain using a standard scoring system (FLACC scale) every few hours after surgery. If the pain score is high (7 or more), the child will receive intravenous paracetamol. Researchers will record how long the pain relief lasts, when the first pain medicine is needed, and the total amount of pain medicine used in the first 24 hours.

The study aims to help doctors choose the most effective and safe method to reduce post-surgery pain in children.

ELIGIBILITY:
Inclusion Criteria:

* Elective infra-umbilical Surgeries
* ASA Status I and II

Exclusion Criteria:

* Chronic systemic illness (cardiovascular, pulmonary or renal disease, hepatic impairment)
* Allergy to local anesthetics
* Coagulation disorder
* Local skin infection
* Neuropathy

Ages: 1 Year to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2025-04-27 (Actual); Primary Completion 2025-07-26 (Actual); Study Completion 2025-07-26 (Actual)

PRIMARY OUTCOMES:
Analgesia Duration | From surgery to 24-hours post operatively
  Duration of post-operative pain free time (hours): time from surgery to FLACC score ≥7 needing rescue analgesia

OTHER OUTCOMES:
Analgesia Consumption | From surgery to 24-hours post operatively
  Total amount (milligrams) of paracetamol consumed

CONTACTS AND LOCATIONS:
Overall Officials: Syed A Abbas Naqvi, FCPS, Study Chair — Allama Iqbal Teaching Hospital Dera Ghazi Khan
Locations (1):
- Allama Iqbal Teaching Hospital, Dera Ghazi Khan, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Saadawy I, Boker A, Elshahawy MA, Almazrooa A, Melibary S, Abdellatif AA, Afifi W. Effect of dexmedetomidine on the characteristics of bupivacaine in a caudal block in pediatrics. Acta Anaesthesiol Scand. 2009 Feb;53(2):251-6. doi: 10.1111/j.1399-6576.2008.01818.x. Epub 2008 Dec 6. PMID 19076110
- [Background] Goyal V, Kubre J, Radhakrishnan K. Dexmedetomidine as an adjuvant to bupivacaine in caudal analgesia in children. Anesth Essays Res. 2016 May-Aug;10(2):227-32. doi: 10.4103/0259-1162.174468. PMID 27212752